CLINICAL TRIAL: NCT02120196
Title: Comparative Study of Rifaximin Versus Norfloxacin in the Secondary Prophylaxis of Spontaneous Bacterial Peritonitis
Acronym: SBP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Dr, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Asem Ahmed Elfert
Record Dates: First submitted 2014-04-07; First posted 2014-04-22 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Spontaneous Bacterial Peritonitis; Ascites; Liver Cirrhosis
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — Rifaximin; Norfloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rifaximin (Experimental): Arm 1: 109 patients will be treated with 1200 mg of rifaximin daily for 6 months.
  Interventions: Drug: Rifaximin
- norfloxacin (Active Comparator): Arm 2: 109 patients will be treated with 400 mg of norfloxacin daily for 6 months.
  Interventions: Drug: Norfloxacin

INTERVENTIONS:
Drug: Rifaximin — rifaximin 1200 mg daily versus norfloxacin 400 mg once daily
  Other Names: Gastrobiotic, Trencedia
  Arms: rifaximin
Drug: Norfloxacin — FDA approved:400mg once daily
  Other Names: Epinor
  Arms: norfloxacin

SUMMARY:
The aim of the study is to compare the effectiveness of rifaximin versus norfloxacin for secondary prevention of spontaneous bacterial peritonitis in patients with liver cirrhosis and ascites.

DETAILED DESCRIPTION:
This study will be carried out on 100 patients with liver cirrhosis and ascites who will be enrolled from Tanta University, Tropical Medicine Department in the period between January 2014 to 6 months. The selected patients will be randomly assigned to receive 400 mg of norfloxacin daily or 1200 mg of rifaximin daily and will be classified into two groups :

Group 1 : 50 patients will be treated with 1200 mg of rifaximin daily. Group 2 : 50 patients will be treated with 400 mg of norfloxacin daily.

ELIGIBILITY:
Inclusion Criteria:

* Previous episode of SBP
* Total protein in the ascitic fluid below or equal to 1.5 g/dL

Exclusion Criteria:

* Allergy to quinolones
* Antibiotic therapy in the 2 weeks preceding inclusion
* Recent ( within the previous 2 weeks) episode of digestive hemorrhage
* Hepatocellular carcinoma or other neoplasias able to shorten life expectancy
* Pregnant and lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recurrence of SBP | 6 months
  The total number of paper of participitants with recurrence of SBP

CONTACTS AND LOCATIONS:
Overall Officials: Asem A Elfert, Principal Investigator — TUH
Locations (1):
- Tanta university hospital, Tanta, Egypt